CLINICAL TRIAL: NCT03928262
Title: A Phase 1, Randomized, Single-blind Study to Assess the Safety, Tolerability, and Pharmacokinetics of Benralizumab Administered as Single Subcutaneous Dose in Healthy Chinese Subjects
Brief Title: Pharmacokinetic Study of Benralizumab in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00034
Record Dates: First submitted 2019-01-28; First posted 2019-04-26 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Safety; Tolerability; Benralizumab; Healthy Chinese subjects
MeSH Terms: interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: 36 healthy Chinese male and female subjects randomized in a 1:1:1 ratio to receive a single SC administration of benralizumab, Treatment 1, Treatment 2 and Treatment 3 (12 subjects per group). Each subject will participate in only 1 treatment group.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Benralizumab - Subcutaneous administration of Dose 1 (Experimental): Benralizumab single dose administration subcutaneously
  Interventions: Biological: Benralizumab
- Benralizumab - Subcutaneous administration of Dose 2 (Experimental): Benralizumab single dose administration subcutaneously
  Interventions: Biological: Benralizumab
- Benralizumab - Subcutaneous administration of Dose 3 (Experimental): Benralizumab single dose administration subcutaneously
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Treatment 1: Benralizumab single dose, Treatment 2: Benralizumab single dose and Treatment 3: Benralizumab single dose subcutaneously administration on 36 healthy Chinese male and female subjects in 1:1:1 ratio.

SUMMARY:
This is a Phase 1, randomized, single-blind study in healthy Chinese subjects at single dose administration of benralizumab: Treatment 1, Treatment 2 and Treatment 3. The study design allows an assessment of 3 doses with safety monitoring and PK sampling to evaluate the safety, tolerability and PK profile of benralizumab.

DETAILED DESCRIPTION:
This study will be conducted at 1 study center in Hong Kong. Approximately 36 healthy Chinese male and female subjects, aged 18 to 45 inclusive, will be randomized in a 1:1:1 ratio to receive a single SC administration of benralizumab: Treatment 1, Treatment 2 and Treatment 3 (12 subjects per group). Each subject will participate in only 1 treatment group. Approximately 8-12 evaluable subjects in each group that met specific non-compartmental analysis (NCA) criteria are required to ensure eligible AUC0-∞ calculation. The total length of the study for each subject is up to 117 days (28 days of screening and 85+/- 4 days of further study visits).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to give written informed consent by signing an IRB/IEC approved Informed Consent Form (ICF) and follow the restrictions and procedures outlined for the study.
2. Healthy adult males or females as determined by medical history, physical examination, and laboratory tests. Subjects age between 18 to 45 years old (inclusive) at the time of signing informed consent. Subject is a Han Chinese who were born in China (including Hong Kong) with Han Chinese parents and grandparents who were born in China (including Hong Kong)
3. Have a body mass index (BMI) between 19 and 24 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg.
4. Medically healthy subjects with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination). Haemoglobin must be greater than the lower limit of normal. A 12-lead ECG with QTc >340 msec and <450 msec.
5. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test prior to administration of the IP and use an effective form of birth control (confirmed by the Investigator or designee). Highly effective forms of birth control include: true sexual abstinence, a vasectomised sexual partner, Implanon, female sterilization by tubal occlusion, any effective IUD Intrauterine device/IUS Ievonorgestrel Intrauterine system, Depo-Provera™ injections, oral contraceptive, and Evra Patch ™ or Nuvaring™. WOCBP must agree to use an effective method of birth control, as defined above, from enrolment, throughout the study duration and within 16 weeks (5 half-lives or longer) after the dosing and have negative serum or urine pregnancy test result on Visit 1 and Visit 2.
6. Women of non-childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
7. Male subjects should be willing to use condoms, in association with another method of contraception, from the day of the first dosing until 16 weeks (5 half-lives or longer) after the dosing.

Exclusion Criteria:

1. Any subject with a history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorder that is capable of altering the metabolism or elimination of drugs or that constitutes a risk factor when taking the study medication.
2. Any subject with a documented history of disorders of the immune system at any time.
3. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with or has failed to respond to standard of care therapy.
4. Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than 1 year prior to Visit 1.
5. Any subject with a clinically significant relevant deviation from normal in physical examination, electrocardiography, or clinical laboratory tests, as determined by the Principal Investigator.
6. Any clinical significant findings off Chest x-rays or CT image. If a chest X-ray or CT has not been performed within 6 months prior to screening visit, a chest X-ray must be performed before the IP administration.
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > the upper limit of normal (ULN).
8. Positive result on screening for serum hepatitis B surface antigen, or hepatitis C antibody. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
9. Any subject with any condition resulting in an increased eosinophil count at screening.
10. Any condition requiring the regular use of any medication.
11. Any subject requiring a prescription medication, other than contraceptives. Subjects taking nonprescription medications must be willing and able to refrain from their use during the inpatient period of the study.
12. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, systemic corticosteroid for condition other than short course for nasal polyps, or any experimental anti-inflammatory therapy) within 3 months prior to the date informed consent is obtained, and during the study period.
13. Receipt of any marketed or investigational biologic (monoclonal or polyclonal antibody) within 4 months or 5 half-lives prior to the date informed consent, is obtained, whichever is longer, and during the study period. E.g. Previous receipt of mepolizumab, reslizumab, dupilumab, or benralizumab.
14. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
15. Receipt of live attenuated vaccines 30 days prior to the date of informed consent.
16. Any subject with known sensitivity to any constituent of benralizumab or any other IL-5 receptor antagonist. History of anaphylaxis to any biologic therapy.
17. Any subject who has participated in any other study of an IP within either 30 days or 5 half-lives (if known) prior to Visit 1, whichever is longer.
18. Current evidence of drug abuse or history of drug abuse within 1 year of randomization, and/or positive results of drug screen and alcohol test at screening and at Day -1.
19. Subjects who have an average weekly alcohol intake that exceeds 21 units per week or subjects unwilling to stop alcohol consumption for the duration of the study (1 unit=12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
20. Smoker of more than 5 cigarettes/day or equivalent use of nicotine products during the previous 3 months from the day of screening.
21. Currently pregnant, breastfeeding or lactating women.
22. Any subject who plans to undergo elective surgery within 4 weeks before Visit 3 (Day 1) through the end of the study (Day 85).
23. Any subject who has donated blood or in any other way had a loss of blood volume greater than 400 mL within 30 days before beginning the study IP administration.
24. Any subject who is unwilling to reside in the clinic during the study period or is unwilling to cooperate fully with the Principal Investigator or designee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse events (AEs) and serious adverse events (SAEs) | Day (-1) to Day 85
  The number and percentage of subjects with treatment-emergent AE/SAE/AE by severity/drug-related AE/drug-related SAE/death in each dose level group and overall. AE/SAE will be displayed by MedDRA SOC and/or PT.
Safety as determined by abnormality in haematology | Day (-1) to Day 85
  Measurement of red blood cell count, white blood cell count, haemoglobin and platelets
Safety as determined by abnormality in clinical chemistry | Day (-1) to Day 85
  Measurement of kidney function (e.g.urea ,creatinine, Uric acid), liver function(ALP, ALT, AST, albumin, total bilirubin), lipid profile(total cholesterol, triglycerides), potassium.
Safety as determined by abnormality in urinalysis | Day (-1) to Day 85
  Measurement of glucose, ketones, leukocytes, blood and protein
Safety as determined by evaluation of blood pressure in mmHg | Day (-1) to Day 85
  Measurement of blood pressure (systolic and diastolic in mmHg)
Safety as determined by evaluation of Pulse rate in beats per minute | Day (-1) to Day 85
  Measurement of Pulse rate in beats per minute
Safety as determined by evaluation of body temperature in degree Celsius | Day (-1) to Day 85
  Measurement of body temperature in degree Celsius
Safety as determined by analysis of 12-lead ECG variables: heart rate (beats per minute) | Day (-1) to Day 85
  The ECG variables will be summarized by absolute value at each visit by treatment group, together with the corresponding changes from baseline.
Safety as determined by analysis of 12-lead ECG variables: PR, QRS, QT and QTcF (milliseconds) | Day (-1) to Day 85
  The ECG variables will be summarized by absolute value at each visit by treatment group, together with the corresponding changes from baseline.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85
  To assess the Pharmacokinetic profile of Subcutaneously administration of benralizumab in healthy Chinese subjects.
Time to maximum observed concentration (tmax) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration of benralizumab in healthy Chinese subjects.
Area under the concentration-time curve from 0 to the last measurable time point (AUC0-t) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration benralizumab in healthy Chinese subjects.
Area under the concentration-time curve from 0 to infinity (AUC0-∞) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration benralizumab in healthy Chinese subjects.
Apparent clearance (CL/F) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration benralizumab in healthy Chinese subjects.
Apparent volume of distribution at terminal phase (Vz/F) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration benralizumab in healthy Chinese subjects.
Time for concentration to decrease by 50% (concentration half-life) (t1/2) | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 2, Day 4, Day 5, Day 6, Day 8, Day 15, Day 29, Day 43, Day 57 and Day 85.
  To assess the Pharmacokinetic profile of subcutaneously administration benralizumab in healthy Chinese subjects.
Anti-drug antibody (ADA) as determined by evaluation of ADA positive percentage and ADA negative percentage | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 29, Day 57 and Day 85.
  To assess the immunogenicity of benralizumab.
All ADA positive samples will be tested for neutralizing antibodies (nAb). nAb as determined by evaluation of nAb positive percentage | Blood samples will be collected from Day 1 (1 hour prior to administration of IP) and on Day 29, Day 57 and Day 85.
  To assess the immunogenicity of benralizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang Tommy Cheung, MBBS, Principal Investigator — HKU Phase 1 Clinical Trials Centre, 2/F, Block K, Queen Mary Hospital, 102 Pokfulam Road, Hong Kong
Locations (1):
- Research Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No